CLINICAL TRIAL: NCT05095298
Title: Reactogenicity and Immunogenicity of Third Dose Vaccine Booster Following Two Doses of Inactivated Vaccines
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director, Huashan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BOOST
Record Dates: First submitted 2021-10-02; First posted 2021-10-27 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Participants volunteered not to receive the third dose of vaccine, and agreed to be followed-up for 1 year
- Inactivated Vaccine Group (Experimental): Participants volunteered to receive the third dose of inactivated vaccine
  Interventions: Drug: Vaccine, COVID19
- Recombinant subunit protein vaccine (Experimental): Participants volunteered to receive the third dose of subunit protein vaccine
  Interventions: Drug: Vaccine, COVID19
- mRNA vaccine Group (Experimental): Participants volunteered to receive the third dose of mRNA vaccine ( To be enrolled, the vaccine has not been approved in China)
  Interventions: Drug: Vaccine, COVID19

INTERVENTIONS:
Drug: Vaccine, COVID19 — It is a prospective open-labeled study, We intended to recruit the participants who completed 2 doses of inactivated COVID-19 vaccine 4-8 months before, and volunteered to receive the third dose of vaccine (inactivated vaccine, recombinant subunit protein vaccine or mRNA vaccine) into the experimental group, and the participants who completed 2 doses of inactivated COVID-19 vaccine 4-8 months before without a third dose of vaccination plan into the control group. Participants in the experimental group received the third dose of SARS-CoV-2 vaccination at baseline, and participants in the control group received no intervention. Each subject will be followed up for one year after enrollment, and neutralizing antibodies and total antibodies will be tested at the specified time points, as well as the records of adverse events and adverse reactions.
  Arms: Inactivated Vaccine Group; Recombinant subunit protein vaccine; mRNA vaccine Group

SUMMARY:
It is a prospective open-labeled study, We intended to recruit the participants who completed 2 doses of inactivated COVID-19 vaccine 4-8 months before, and volunteered to receive the third dose of vaccine (inactivated vaccine, recombinant subunit protein vaccine or mRNA vaccine) into the experimental group, and the participants who completed 2 doses of inactivated COVID-19 vaccine 4-8 months before without a third dose of vaccination plan into the control group. Participants in the experimental group received the third dose of SARS-CoV-2 vaccination at baseline, and participants in the control group received no intervention. Each subject will be followed up for one year after enrollment, and neutralizing antibodies and total antibodies will be tested at the specified time points, as well as the records of adverse events and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Through asking medical history and physical examination, the investigator judged that the health condition is good: the chronic disease is stable and there is no change within 3 months of medication;
* has been completed 2 doses of Covid-19 Inactivated vaccine 4-8 months ago;
* Female participants of childbearing age who were not breast-feeding or pregnant (negative blood pregnancy test), and had no family planning in the first 3 months after enrollment and took effective contraceptive measures. Take effective contraceptive measures within 2 weeks before inclusion;
* Volunteered to receive the third dose of vaccine.And during the entire follow-up research period, be able and willing to complete the entire prescribed research plan; Have the ability to self-understand research procedures, informed consent & voluntarily sign informed consent, and be able to comply with the requirements of the plan

Exclusion Criteria:

* RT-qPCR detects active SARS-Cov-2 infection;
* a history of COVID-19, SARS, MERS infection (self-report, on-site inquiry);
* a high-risk factor for COVID-19 infection:
* a history of close contact with people infected with the new coronavirus, a history of living in high-risk areas, and a history of contact with patients with fever or respiratory symptoms in high-risk areas or abroad.
* Fever, dry cough, fatigue, nasal congestion, runny nose, sore throat, myalgia, diarrhea, shortness of breath, dyspnea, etc. 7 days before enrollment;
* receiving COVID-19 booster vaccination;
* allergic to the active ingredients of the SARS-CoV-2 vaccine, any of the inactive ingredients, the substances used in the production process, or those who have had allergies during previous vaccination of similar vaccines;
* those who have had severe allergic reactions to vaccines in the past (such as acute allergic reactions, angioedema, respiratory Difficulties, urticaria, angioedema or abdominal pain);
* body temperature >37.0℃ before vaccination;
* blood pregnancy test positive;
* with uncontrolled epilepsy and other serious neurological diseases (such as transmissive myelitis, Guillain-Barre syndrome) , Demyelinating diseases, etc.), or have a history or family history of encephalopathy or mental disease;
* severe liver and kidney disease, uncontrollable hypertension (systolic blood pressure ≥180 mmHg, diastolic blood pressure ≥100 mmHg), diabetic complications, Malignant tumors, various acute diseases or acute attacks of chronic diseases;
* diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* receiving anti-tuberculosis treatment;
* a history of coagulopathy ( Such as coagulation factor deficiency, coagulation disease) within 3 months of subjects receiving immunotherapy or inhibitor therapy (continuous oral or infusion for more than 14 days), or after 3 months of hormone therapy, the average daily dose is ≥20mg/day (Prednisone);
* Receiving live attenuated vaccine within 1 month before this vaccination, other vaccines within 14 days before this vaccination;
* Receiving other research drugs within 3 months before vaccination; participating in other research vaccines Or subjects in clinical trials of research drugs;
* other conditions that the investigator judges are not suitable for this clinical trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of Third Dose Vaccine Booster Following Two Doses of Inactivated Vaccines | Day 28
  Observe the 28th day of the subjects' pseudovirus neutralizing antibody geometric mean titers (GMTs) and mean geometric titers fold growth (GMFR) changes
Reactogenicity of Third Dose Vaccine Booster Following Two Doses of Inactivated Vaccines | Day 28
  All solicited and non-solicited adverse events within 28 days.

SECONDARY OUTCOMES:
The seropositive rate of neutralizing antibodies | 3 days/14 days/28days/45days/60 days/90 days/180 days/365 days
  The seropositive rate of neutralizing antibodies after third vaccination shots
GMT of neutralizing antibodies | 3 days/14 days/28days/45days/60 days/90 days/180 days/365 days
  GMT of neutralizing antibodies after third vaccination shots
GMFR of neutralizing antibodies | 3 days/14 days/28days/45days/60 days/90 days/180 days/365 days
  GMFR of neutralizing antibodies after third vaccination shots
severe adverse events and adverse events of special interest | up to 1 year
  severe adverse events and adverse events of special interest

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Huashan Hospital affiliated to Fudan University, Shanghai, Jingan
  - Beijing Ditan Hospital Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Undecided